CLINICAL TRIAL: NCT04148781
Title: The Effect of Fampridine-SR on Visual Function in Poorly Recovered Optic Neuritis in Persons With MS
Brief Title: Fampridine-SR and Optic Neuritis Recovery
Acronym: FAMP-ON
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Courtney Casserly (Other)
Responsible Party: Sponsor-Investigator, Courtney Casserly, Neurologist, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113427
Record Dates: First submitted 2019-09-11; First posted 2019-11-04 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Optic Neuritis
Keywords: Multiple sclerosis; Optic Neuritis; Fampyra
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fampridine-SR (Experimental): Fampridine-SR 10 mg Orally Twice Daily for 8 weeks.
  Interventions: Drug: Fampridine SR

INTERVENTIONS:
Drug: Fampridine SR — Fampridine-SR 10 mg twice daily for 8 weeks

SUMMARY:
Optic Neuritis (ON) is a condition that occurs in approximately 50% of individuals with relapse remitting MS, and is the presenting event in 15-20% of patients who go on to develop MS. These ON events present with a decline in vision over several days with painful eye movements. The purpose of this study is to collect pilot data on the effect of Fampridine-SR on the recovery of visual function after demyelinating optic neuritis.Our team evaluated a person with ON who had incomplete recovery which was quite bothersome to her. After a one-month treatment course Fampridine SR,her visual functioning improved. Based on this case, we present a unique opportunity to evaluate the potential benefit of Fampridine-SR as a potential treatment for persons who do not fully recover from acute ON.

DETAILED DESCRIPTION:
Optic Neuritis (ON) is a condition that occurs in approximately 50% of individuals with relapse remitting MS, and is the presenting event in 15-20% of patients who go on to develop MS. ON usually presents with a decline in vision over several days to weeks with painful eye movements.

Fampridine-SR is currently a Health Canada approved medication to treat walking impairment in persons with MS. Some small studies in the past have shown that Fampridine-SR may also have positive effects on visual functioning in those experiencing ON.

This study will aim to assess the effect of taking Fampridine-SR for 8 weeks in 20 MS patients with unresolved optic neuritis on measures of visual functioning, and to determine the best measures to use in a future large scale study. The results of this study will also be used to estimate how many participants we will need in the future large scale study.

ELIGIBILITY:
Inclusion Criteria:

* Have an MS diagnosis, any type
* Had an acute optic neuritis without full recovery which occurred ≥ one year ago
* Have a visual acuity in the affected of eye of ≥ 20/40 or

  1. Or ≥20 ms difference in VEP between eyes
  2. Or ≥ 120 ms VEP in the affected eye
* Have not received corticosteroids in the last thirty (30) days
* Medications that could potentially affect the VEP P100 amplitude or may cause drowsiness/difficulty with visual fixation are allowed if there has been no change in dose within 30 days of study enrollment or anytime during the study. These medications include:

  1. Benzodiazepines other than every night at bedtime
  2. Opioid and opiates other than every night at bedtime
  3. Cannabinoid products other than every night at bedtime
* Have given written informed consent prior to any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care

Exclusion Criteria:

* Have another medical condition that could affect the visual outcomes, such as, but not limited to, diabetes retinopathy, glaucoma, cataracts, previous ocular trauma, amblyopia, and optic neuropathy not due to a demyelinating lesion
* Creatinine clearance ≤ 80 mL/min
* Has a history of seizures, with the exception of febrile seizure as an infant
* Taking a medicinal product that is an inhibitor of Organic Cation Transporter 2 (OCT-2)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Evoked Potentials | Measured at baseline, week 8, and week 12
  Visual evoked potentials (VEPs) measure the occipital cortical response to visual stimuli and are used to detect visual abnormalities. VEPs will be measured at multiple time points to assess any changes in VEPs over the duration of the study.
Change in Visual Acuity | Measured at baseline, week 8, and week 12
  Change in visual acuity will be assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts and standard protocol as it the gold standard for ophthalmology clinical trials using visual acuity as an outcome. Visual acuity will be measured at multiple time points to assess any changes over the duration of the study.
Change in Contrast Sensitivity | Measured at baseline, week 8, and week 12
  Contrast sensitivity or low contrast visual acuity (LCVA) has been found to be a sensitive measure of visual function in demyelinating lesions when focusing on recovery, even in patients with high contrast visual acuity. Contrast sensitivity will be measured at multiple time points to assess any changes over the duration of the study.
Change in Colour Vision | Measured at baseline, week 8, and week 12
  Colour vision is frequently affected in optic neuritis and unlikely to fully recover We will use Ishihara colour plates, a common test to assess colour vision. Colour vision will be measured at multiple time points to assess any changes over the duration of the study.
Change in Visual Fields | Measured at baseline, week 8, and week 12
  Measures of central visual function are important in the evaluation of optic neuritis, because most cases of optic neuritis affect central vision and therefore decrease quality of life. Visual fields will be measured at multiple time points to assess any changes over the duration of the study.
Optical Coherence Tomography | Measured at baseline.
  Optical coherence tomography (OCT) is now a ubiquitous technology in the world of MS research, and is an excellent means of imaging the layers of the retina.
Change in 10-Item Neuro-Ophthalmic Supplement total scores | Measured at baseline, week 8, and week 12
  The 10-Item Neuro-Ophthalmic Supplement (NOS-10) has been developed to capture patient-reported outcomes related to visual dysfunction in patients with visual disorders. Total scores will be collected (range 1 to 52). Scores on the NOS-10 will be measured at multiple time points to assess any changes over the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada